CLINICAL TRIAL: NCT00804791
Title: Residence Time Evaluation of Marketed OTC Ophthalmic Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M-08-11
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: dry eye; autofluorescence; residence time
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane (Active Comparator): One drop dispensed into each eye
  Interventions: Other: Systane Ultra Lubricant Eye Drops
- Unisol (Active Comparator): One drop dispensed into each eye
  Interventions: Other: Unisol 4 Saline Solution

INTERVENTIONS:
Other: Systane Ultra Lubricant Eye Drops — artificial tears solution for lubricating the cornea
  Arms: Systane
Other: Unisol 4 Saline Solution — saline solution for irrigating the cornea
  Arms: Unisol

SUMMARY:
The objective of this study is to measure ocular surface residence time (in minutes) of two marketed OTC ophthalmic products in dry eye patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and HIPAA read, signed and dated before conducting any procedures.
* Adult volunteers diagnosed with mild to moderate dry eye. Criteria for diagnosis must include 2 of the 3 following characteristics: composite symptom score > or = to 5 on modified Schein questionnaire; NaFl TFBUT < or = to 7 seconds in either eye; or NaFl corneal staining sum score > or = to 3 (using 0-15 point grading system).
* Able and willing to follow study instructions. 4) Best-corrected V.A. of 0.6 logMAR or better OU.

Exclusion Criteria:

* History or evidence of ocular or intraocular surgery in either eye w/i the past 6 months.
* History or evidence of serious ocular trauma in either eye w/i the past 6 months.
* History of intolerance or hypersensitivity to any component of the study medications.
* History or evidence of epithelial herpes simplex keratitis, vaccinia, active or recent varicella viral disease of the cornea and/or conjunctiva and/or eyelids, mycobacterial infection of the eye, and/or fungal disease of the eye.
* Use of concomitant topical ocular medications during the study period.
* Patients using systemic medications that may contribute to dry eye may not be enrolled unless they have been on a stable dosing regimen for a minimum of 30 days prior to Visit 1, and the dosing regimen must remain stable throughout the study period.
* Ocular conditions such as conjunctival infections, iritis, or any other ocular condition that may preclude the safe admininstration of the test article.
* Individuals unwilling to d/c contact lens wear during the study period. CL wear must have been d/c at least one week prior to Visit 1.
* Participation in an investigational drug or device study w/i 30 days of entering this study.
* Additionally, any subject may be declared ineligible for a valid medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Residence Time | After 8 minutes, then every 2 minutes
  Ocular surface residence time is the time for fluorescent intensity of the cornea to return to baseline measurement after installation of test article.